CLINICAL TRIAL: NCT02104505
Title: Effect of Gamma Tocopherol Enriched Supplementation on Response to Inhaled LPS
Acronym: Vitalps
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Purdue University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-1605; R01ES023349 (NIH)
Record Dates: First submitted 2014-03-24; First posted 2014-04-04 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-09

CONDITIONS: Mild, Allergic Asthma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — gamma-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 700 mg Gamma Tocopherol daily x 14days (Active Comparator): Gamma Tocopherol supplement
  Interventions: Drug: Gamma Tocopherol 700 mg capsules,
- Placebo (Placebo Comparator): Safflower oil capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gamma Tocopherol 700 mg capsules, — 2 capsules daily
  Arms: 700 mg Gamma Tocopherol daily x 14days
Drug: Placebo — Safflower oil capsules
  Arms: Placebo

SUMMARY:
To test the hypothesis that gamma tocopherol (vitamin E) supplement inhibits endotoxin induced airways inflammation in allergic asthmatics

DETAILED DESCRIPTION:
BACKGROUND:

Allergic asthma (AA) is the most commonly encountered respiratory disease in children and adults in the United States and is a leading cause of morbidity worldwide. Among the most disruptive expressions of disease in AA is acute asthma exacerbation. The Center for Disease Control lists ambient air pollutants and environmental tobacco smoke as among the most common triggers for acute asthma exacerbation. Ozone (O3) is the most commonly encountered ambient air pollutant in the US. Endotoxin (or lipopolysaccharide or LPS) is a component of bioaerosols found in both the indoor and outdoor environment, is a component of tobacco smoke, and is increased in indoor settings where smokers live. LPS is also a component of coarse and fine mode particle matter air pollution.

OXIDATIVE STRESS AND ASTHMA:

Increased oxidative stress and decreased antioxidant capability have been observed in asthmatics. These pollutants are pro-inflammatory and are associated with increased oxidative stress, which would exacerbate reactive oxygen and reactive nitrogen species (ROS and RNS)-induced injury in asthmatics. O3 injures epithelial cells, releasing secondary mediators which activate inflammatory cells, in part by ligation of Toll-Like Receptor 4 (TLR4), the primary receptor for LPS. TLR4 activation of inflammatory cells activates Nuclear Factor-kB (NF-kB) and induces oxidative stress. O3 and LPS has been associated with exacerbation of asthma, and we have reported that O3 and LPS augments allergic airway inflammation in allergic asthmatics (AA). Development of interventions to mitigate these responses will greatly decrease disease morbidity.

Given the role that oxidants play in the pathophysiology of asthma exacerbation, defects in antioxidant levels would increase risk for acute asthma exacerbation. Nutritional deficiencies in vitamin E, ascorbate and selenium have been linked to asthma severity, and asthmatics have decreased antioxidant levels in airway fluid. We and others have shown that vitamins C and E are decreased in airway fluids of asthmatics. Additionally, genetic factors may increase risk for oxidant induced exacerbation of asthma. Many investigators have reported that persons who are homozygous for the null polymorphism of the Glutathione-S-Transferase Mu1 (GSTM1) gene and unable to produce GSTM1 protein (the GSTM1 null genotype) have increased risk of acute pollutant-induced exacerbation of asthma. We have shown in healthy volunteers that the GSTM1 null genotype is associated with increased inflammatory response to O3, with no impact on the nociceptive response to this pollutant. We have also shown that GSTM1 null volunteers have enhanced airway and systemic inflammation following LPS challenge.

Others have shown that the GSTM1 null genotype is associated with increased response to secondhand tobacco smoke, diesel exhaust, and other particulate matter components. Romieu et al demonstrated that children with asthma in Mexico City were had increases susceptibility to O3-induced exacerbations if they had the GSTM1 null genotype. This group also found that GSTM1 null AAs selectively benefited from antioxidant intervention. The GSTM1 null genotype is found in 20-40% of the population, and may be overrepresented in allergic populations. Taken together, these observations show that the sizable GSTM1 null population is at risk for pollutant-induced airway disease, and that antioxidant intervention targeting the action of ROS and RNS will benefit asthmatics and especially GSTM1 null asthmatics.

ANTIOXIDANTS AND ASTHMA:

A non-exclusive list of proposed antioxidants includes radical scavengers such as ascorbate, a-tocopherol (aT), y-tocopherol (yT) or inducers of the antioxidant gene response element transcription factor NRF2, which activate NRF2 with subsequent broad upregulation of acute phase II and antioxidant proteins. These agents are available in naturally occurring foods and as nutritional supplements. A number of animal, cell culture and epidemiological studies support the idea that antioxidant supplementation is useful in allergic airway disease. However, despite these studies and widespread public and scientific enthusiasm regarding use of such agents in asthmatics, there are scant human data to support or refute the use of such interventions for either acute or chronic allergic airways disease. It is crucial that adequate, well-designed human studies assess the role of antioxidants for allergic asthma to either confirm their efficacy, or refute claims that these are effective, safe and low cost interventions for allergic disease.

GAMMA TOCOPHEROL AND ASTHMA:

Gamma tocopherol has both radical scavenging and anti-inflammatory actions which may play important roles in decreasing pollutant-induced and allergic injury to the airway.

Like other isoforms of vitamin E, yT is a potent ROS scavenger and is also a powerful nucleophile that traps electrophiles such as peroxynitrite in lipophilic compartments. One mechanism by which y-T is cytoprotective is scavenging of RNS at the un-substituted C-5 position on the hydroxy-chroman ring of y-T to form 5-NO-y-tocopherol (5-NO-yT). Overall, vitamin E provides general protection of DNA, lipids and proteins from radical stress. An example of such protection is shown in rodent studies of prostate cancer in which intake of yT is associated with decreased DNA methylation of CpG rich regions of the NRF2. NRF2 is a master regulator of numerous cytoprotective antioxidant enzymes.

Supplementation with yT also prevents protein nitration and attenuates loss of plasma vitamin C in plasma in a rodent peritonitis model of inflammation. Our group has also shown that yT inhibits cyclo-oxygenase-2 (COX-2) and 5-lipoxygenase (5-LO) in LPS-stimulated macrophages and interleukin (IL)-1b stimulated epithelial cells. These actions are mediated primarily by the yT metabolite 2, 7, 8-trimethyl-2S-(.-carboxyethyl)-6-hydroxychroman (y-CEHC) which requires hydroxylation of the y-methyl group of yT by cytochrome P450 (CYP450). In carrageenan- induced inflammation in male Wistar rats, yT decreases prostaglandin (PGE2) and leukotriene (LTB4) production, suggesting that 5-LO-mediated production of leukotrienes may also be inhibited by yT. Tocopherols, including yT, also modulate gene expression of a number of inflammatory genes. Thus, yT and other tocopherols decrease production of a number of pro-inflammatory cytokines at the transcriptional level.

In animals, we have also shown that gamma tocopherol reduces baseline eosinophilia in the airway. In our early phase I studies of gamma tocopherol-enriched mixed tocopherols (gT-mT) we have shown that gT-mT inhibits monocyte induced cytokine production, decreases baseline nitrosative stress, and inhibits LPS eosinophil and neutrophil influx in healthy volunteers.

SUMMARY:

There is widespread opinion that antioxidant nutrients like gamma tocopherol ( yT, a form of Vitamin E) are an untapped and inexpensive intervention for environmentally triggered acute asthma. However, there is a crucial gap in evidence-based support of such interventions in asthma. A lack of coordinated research assessing specific antioxidant regimens from preclinical, phase I and phase II studies impedes development of phase III antioxidant trials in asthmatic populations. It is also unclear which physiological endpoints are most relevant in such studies. This project focuses on phase II studies of yT in AA based on our preclinical and phase I studies. For this protocol we will be testing the hypothesis that a gamma tocopherol supplement will baseline eosinophil numbers in airway sputa of asthmatics (specific aims 1) and (specific aim 2) inhibit LPS induced airway inflammation in mild allergic asthmatics.

The investigators will also do an exploratory assessment of the specific impact of the GSTM1 null genotype on response to LPS and effect of gamma tocopherol enriched supplementation on this response.

If gamma tocopherol decreases LPS-induced response in asthmatics, this would provide proof of concept that this agent would be a useful intervention for asthma, confirming teh need for a phase III study of gamma tocopherol enriched supplements as a treatment for asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 of both genders
2. Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
3. History of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician diagnosed asthma.
4. Positive methacholine test. A positive test is defined as a provocative concentration of methacholine of 10 mg/ml or less producing a 20% fall in Forced Expiratory Volume in 1 second (FEV1) (PC20 methacholine) by the method used in a separate screening protocol.
5. FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .70 (without use of bronchodilating medications for 12 hours or long acting beta agonists for 24 hours), consistent with lung function of persons with no more than mild episodic or mild persistent asthma.
6. Allergic sensitization to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive immediate skin test response.
7. Symptom Score (this will be submitted as an attachment) no greater than 16 (out of a possible 24) for total symptom score with a value no greater than 3 for any one score. No more than one score may be greater or equal than 3.
8. subjects must be willing to avoid caffeine for 12 hours prior to all visits.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency, history of tuberculosis
2. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months
3. Moderate or Severe asthma
4. Exacerbation of asthma more than 2x/week which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
5. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current National Heart, Lung and Blood Institute (NHLBI) guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
6. Viral upper respiratory tract infection within 2 weeks of challenge.
7. Any acute infection requiring antibiotics within 2 weeks of exposure or fever of unknown origin within 2 weeks of challenge.
8. Severe asthma
9. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
10. Medications which may impact the results of the Clinical Center Reference Endotoxin (CCRE) exposure, interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents)
11. Any history of smoking in the year prior to study enrollment; lifetime smoking history > 10 pack years
12. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma
13. Allergy/sensitivity to study drugs, including E coli, or their formulations.
14. Known hypersensitivity to methacholine or to other parasympathomimetic agents
15. History of intubation for asthma
16. Unwillingness to use reliable contraception if sexually active (Intrauterine device, birth control pills/patch, condoms).
17. Abnormal Prothrombin Time (PT) or Partial Thromboplastin Time (PTT) values at screening or during the treatment period. Normal values will be those published by the clinical lab (Labcorp, INC).
18. Any bleeding disorder
19. Radiation exposure history will be collected. Subjects whose exposure history within the past twelve months would cause them to exceed their annual limits will be excluded.
20. Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Burbank AJ, Duran CG, Pan Y, Burns P, Jones S, Jiang Q, Yang C, Jenkins S, Wells H, Alexis N, Kesimer M, Bennett WD, Zhou H, Peden DB, Hernandez ML. Gamma tocopherol-enriched supplement reduces sputum eosinophilia and endotoxin-induced sputum neutrophilia in volunteers with asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1231-1238.e1. doi: 10.1016/j.jaci.2017.06.029. Epub 2017 Jul 20. PMID 28736267

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no wash out or run-in phase prior to treatment assignment. No enrolled participants were excluded prior to treatment assignment.
Groups:
- Gamma Tocopherol (14 Days) Then Placebo (14 Days): Gamma Tocopherol (2 capsules, each containing 700 mg, daily) x 14 days, washout for minimum 3 weeks, then Safflower oil capsules x 14 days
- Placebo (14 Days) Then Gamma Tocopherol (14 Days): Safflower oil capsules x 14 days, washout for minimum 3 weeks, then Gamma Tocopherol (2 capsules, each containing 700 mg, daily) x 14 days
Period: First Intervention (14 Days)
Arm/Group | Gamma Tocopherol (14 Days) Then Placebo (14 Days) | Placebo (14 Days) Then Gamma Tocopherol (14 Days)
Started | 12 | 11 (one participant withdrew prior to receiving study drug)
Completed | 10 | 8
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — exclusionary condition | 0 | 1
Period: Washout (Minimum 3 Weeks)
Arm/Group | Gamma Tocopherol (14 Days) Then Placebo (14 Days) | Placebo (14 Days) Then Gamma Tocopherol (14 Days)
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Gamma Tocopherol (14 Days) Then Placebo (14 Days) | Placebo (14 Days) Then Gamma Tocopherol (14 Days)
Started | 10 | 8
Completed | 8 | 7
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gamma Tocopherol (14 Days) Then Placebo (14 Days) | Placebo (14 Days) Then Gamma Tocopherol (14 Days) | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23.5 [20 to 42] | 30 [21 to 47] | 26 [20 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23
Atopy [Count of Participants; unit: Participants] | 9 | 8 | 17
Body Mass Index (BMI) [Median (Full Range); unit: kg/m2] | 27.1 [20.5 to 34.8] | 25.2 [20.2 to 41.7] | 26 [20.2 to 41.7]
Forced expiratory volume in 1 second (FEV1) (%predicted) [Median (Full Range); unit: percent predicted] | 102.5 [89 to 109] | 90 [83 to 108] | 97 [83 to 109]

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Change in Sputum Percent Neutrophils (PMN)s Following Inhaled Clinical Center Reference Endotoxin (CCRE) Challenge as Affected by Gamma Tocopherol
Description: In asthmatic individuals, exposure to CCRE is expected to increase PMNs in the sputum. The sputum PMNs were measured at baseline (immediately prior to dosing) and again on day 14 of treatment (approximately 8 hours after the final dose) with placebo or gamma tocopherol. The outcome is to compare the change in PMNs from baseline to post treatment after exposure to CCRE
Time Frame: after 14 days of gamma tocopherol or placebo treatment
Population: Since this study employed a crossover design, only participants who completed both arms of the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: change in percentage of PMNs in sputum
Groups:
- Gamma Tocopherol: Gamma Tocopherol 700 mg capsules,: 2 capsules daily for 14 days
- Placebo: 700 mg Safflower oil capsules; 2 capsules daily for 14 days
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 15 | 15
change in percentage of PMNs in sputum | 11.7 (20.7) | 20.1 (16.5)
Statistical Analysis 1: Comparison: Gamma Tocopherol vs Placebo; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Net) = 0.41, Standard Error of Mean 0.18 — Comparison of change in sputum %PMNs during active treatment vs placebo (crossover design)

2. Secondary Outcome: Chronic Eosinophilic Airway Inflammation as Affected by Gamma Tocopherol
Description: The sputum eosinophils were measured at baseline (immediately prior to dosing) and again after 14 days of treatment (approximately 8 hours after the final dose) with placebo or gamma tocopherol. The outcome is to compare sputum eosinophils per mg before and after gamma tocopherol treatment.
Time Frame: after 14 days of gamma tocopherol or placebo treatment
Population: Since this study employs a crossover design, only participants who completed both arms of the study were included in the final analysis.
Measure: Mean (Standard Deviation); unit: eosinophils per mg sputum
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 15 | 15
eosinophils per mg sputum | 2.6 (4.3) | 9.5 (14.3)
Statistical Analysis 1: Comparison: Gamma Tocopherol vs Placebo; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Net) = 0.64, Standard Error of Mean 0.22

3. Secondary Outcome: Mucociliary Clearance (MCC) Associated With CCRE Challenge as Affected by Gamma Tocopherol
Description: On day 14 of treatment (approximately 6 hours after the final dose) with placebo or gamma tocopherol, a whole lung region of interest (ROI) bordering the right lung was used to estimate (by computer analysis) whole lung retention of inhaled radiolabeled particles. This was performed by measuring the labeled particle counts over a 2 hour period and determining the fraction of initial particle counts remaining. From this data, we determined the percentage of labeled particles cleared from the lung during the 2 hour observation period.
Time Frame: after 14 days of gamma tocopherol or placebo treatment
Population: Due to the crossover design of the study, only participants who completed both arms of the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: % of labeled particles cleared from lung
Groups:
- Gamma Tocopherol: Gamma Tocopherol 700 mg capsules: 2 capsules daily for 14 days
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 15 | 15
% of labeled particles cleared from lung | 20.2 (8) | 16.3 (9.3)
Statistical Analysis 1: Comparison: Gamma Tocopherol vs Placebo; Test type: Superiority; p = 0.6, Mixed Models Analysis; Mean Difference (Net) = -0.32, Standard Error of Mean 0.33

4. Secondary Outcome: Mucociliary Clearance as Affected by Gamma Tocopherol
Description: On day 11 of treatment (approximately 6 hours after the daily dose) with placebo or gamma tocopherol, a whole lung region of interest (ROI) bordering the right lung was used to estimate (by computer analysis) whole lung retention of inhaled radiolabeled particles. This was performed by measuring the labeled particle counts over a 2 hour period and determining the fraction of initial particle counts remaining. From this data, we determined the percentage of labeled particles cleared from the lung during the 2 hour observation period.
Time Frame: after 11 days of gamma tocopherol or placebo treatment
Population: Due to the crossover study design, only participants who completed both arms of the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: % of labeled particles cleared from lung
Arm/Group | Gamma Tocopherol | Placebo
Number analyzed (Participants) | 15 | 15
% of labeled particles cleared from lung | 21.4 (9.7) | 21.4 (6.9)
Statistical Analysis 1: Comparison: Gamma Tocopherol vs Placebo; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mean Difference (Net) = -0.32, Standard Error of Mean 0.33

ADVERSE EVENTS:
Time Frame: 3 months on average
Groups:
- Gamma Tocopherol: Gamma Tocopherol 700 mg capsules; 2 capsules daily for 14 days
Arm/Group | Gamma Tocopherol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 11/17 | 14/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gamma Tocopherol (N=17) | Placebo (N=20)
Headache (Nervous system disorders) | 2 (2) | 1 (2)
Cough during CCRE challenge (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) — Cough observed during CCRE challenge
Diminished sense of taste (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — 5 mm x 5 mm erythematous area underneath the chest patch applied during mucociliary clearance measurement
Vagal response (Cardiac disorders) | 1 (1) | 0 (0) — nausea, lightheadedness, pallor during phlebotomy
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough during sputum induction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of breath during sputum induction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No